CLINICAL TRIAL: NCT04091984
Title: The PROspera Kidney Transplant ACTIVE Rejection Assessment Registry (ProActive)
Acronym: ProActive
Status: Active, not recruiting | Type: Observational
Sponsor: Natera, Inc. (Industry)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Other Study IDs: 18-039-TRP; Pro00037470 (Other: Advarra IRB)
Record Dates: First submitted 2019-09-06; First posted 2019-09-17 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant Rejection
Keywords: donor-derived cfDNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — There are two arms to this study: A prospective arm and a historical control (retrospective arm).
  Each participant in the Prospective arm will have received the commercially available Prospera test.
  Subjects prospectively enrolled and whom consent to "Optional future Research" may have bio-specimens stored for future research.
  The historical arm (retrospective cohort) will not have any bio-specimens collected or stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospera Arm: There is no intervention in this study. Adult patients who have received a kidney allograft from a genetically different donor in the past 2 years including within 60 days and who have been selected by their healthcare provider to receive Prospera dd-cfDNA testing according to their regular interval testing schedule as part of their clinical care will have medical records pertaining to their kidney rejection status collected at each study visit.
  Interventions: Diagnostic Test: Prospera
- Control Arm: The control arm will consist of retrospective data review of cases where a renal allograft from a genetically different donor was performed. Data pertaining to to their kidney rejection status from a minimum of 3 time points per year post allograft (up to 5 years) or until renal allograft failure will be collected.

INTERVENTIONS:
Diagnostic Test: Prospera — No Interventions, this is an observational study.
  Groups: Prospera Arm

SUMMARY:
The ProActive registry is a longitudinal, multi-center study with a prospective arm observing clinical care for patients receiving physician ordered Prospera, an allograft rejection test, and a historical control arm collecting data on cases at the same sites whose kidney allograft rejection status was managed with Serum Creatinine SCr/estimated Glomerular Filtration Rate eGFR. This registry will compare patient management and outcomes in patients who receive Prospera (Prospera arm) to the outcomes of the historical control group (control arm) to determine Prospera's clinical utility. High-risk subjects defined as having a biopsy-demonstrated rejection event or at least one pre-existing Donor Specific Antibody DSA with total Mean Fluorescent Intensity MFI>3000 or a calculated Panel Reactive Antibodies cPRA>70% will be followed for an additional period up to 24 months in both the Prospera arm and historical control arm.

DETAILED DESCRIPTION:
The primary objective is to differentiate the clinical utility of Prospera testing from the use of creatinine testing as measured by the proportion of positive biopsies in post renal allograft patients.

Secondary objectives include:

* To observe the performance of the Prospera assay in detecting AR (repeated validation)
* To evaluate whether Prospera can detect AR earlier and more often than SCr
* To determine whether use of Prospera will significant decrease the rate of overall number of biopsies when compared to the rate of biopsies in the control arm

ELIGIBILITY:
Inclusion Criteria Prospera Arm:

1. 18 years of age or older
2. Renal allograft (kidney transplant) up to 2 years prior to signing informed consent. Newly transplanted patients to receive Prospera testing within 60 days of transplant
3. A genetically different donor (not an identical twin)
4. Selected by a healthcare provider to receive Prospera dd-cfDNA test according to the regular interval testing schedule as part of their practical care
5. Able to read, understand and provide written informed consent
6. Willing and able to comply with the study visit schedule and study requirements

Exclusion Criteria Prospera Arm:

1. Pregnant
2. Routine ongoing testing with another dd-cfDNA or RNA biomarker test after enrollment into the ProActive study. Receipt of another dd-cfDNA test within 30 days of a patient being enrolled in the study.
3. History of another organ transplant (i.e. aside from renal allograph)
4. A serious medical condition that may adversely affect ability to participate in the study (e.g, dementia, current diagnosis of cancer)
5. Previously enrolled in the ProActive Registry, with the exception of a graft failure and a new renal allograft

Inclusion Criteria Control Arm:

1. 18 years of age or older at the time of transplant
2. Had a renal allograft
3. Had a genetically different donor
4. Had a minimum of three evaluations per year during the three years since the renal allograft or until allograft failure

Exclusion Criteria Control Arm:

1. Female patients who were pregnant at any time during the 3-year historical control data collection period
2. Had a transplanted organ other than kidney
3. Received results from a dd-cfDNA test designed to assess renal allograft rejection during the historical control data collection period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 5,000 adult renal allograft participants will be enrolled in this study, and data will be collected from a de-identified cohort of approximately 500 historical control patients who had a renal allograft.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Efficiency of biopsies | 3 years
  The proportion of clinically indicated biopsies that show Active Rejection (AR) will be measured in the Prospera arm and the control arm. Specifically, the proportion of clinically indicated biopsies showing AR in individuals with a positive donor derived-cell free DNA dd-cfDNA test at the time of Bx in the test arm, where Prospera has been integrated into the care paradigm, will be compared against the proportion of clinically indicated biopsies showing AR in the control arm.
Graft function | 3 years
  Graft function in the Prospera arm and control arm will be measured. This will be assessed by examining the average eGFR score (as calculated using serum creatinine Chronic Kidney Disease-EPIdemiology collaboration CKD_EPI equation) at year three in the Prospera arm compared to the average eGFR score determined at year three in the historical control arm.

SECONDARY OUTCOMES:
Evaluate the performance of Prospera | 5 years
  The performance of Prospera to detect AR will be evaluated. The sensitivity, specificity, Positive & Negative Predictive Value of the assay in sub-cohorts of patients will be calculated and compared to the performance of serum creatinine to detect AR in those cohorts.
Evaluate whether Prospera can detect acute rejection earlier than serum creatinine | 3 years
  The grade of rejection observed in biopsies in the Prospera arm will be compared to the historical control arm which used serum creatinine.
Determine if and how Prospera testing impacts patient care | 5 years
  The proportion of Prospera assay results that doctors felt influenced their decisions around management of patients and biopsies will be calculated. This will be analyzed separately for the for-cause and protocol biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bromberg, MD, Principal Investigator — University of Maryland
Locations (55):
- United States (55):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Kidney Disease & Hypertension Centers, Phoenix, Arizona
  - Arizona Kidney Disease & Hypertension Centers, Scottsdale, Arizona
  - Arizona Kidney Disease and Hypertension Centers, Tucson, Arizona
  - Arizona Kidney Disease & Hypertension Centers, Tucson, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - University of California Davis Medical Center, Davis, California
  - University of California, Irvine, Irvine, California
  - Keck School of Medicine USC, Los Angeles, California
  - The Regents of the University of California on behalf of its Los Angeles campus, Los Angeles, California
  - Riverside Community Hospital, Riverside, California
  - California Institute of Renal Research, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Florida Health Sciences Center, Tampa, Florida
  - Cleveland Clinic Florida (Weston), Weston, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - The University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Renal Transplant Associates of New England, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Harper University Hospital, Detroit Medical Center, Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Northwell Health, Inc, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - The Research Institute at Westchester Medical Center, Valhalla, New York
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Toledo, Toledo, Ohio
  - Legacy Research, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Kidney Care Specialists, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - IHC Health Services, Inc, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bromberg JS, Bunnapradist S, Samaniego-Picota M, Anand S, Stites E, Gauthier P, Demko Z, Prewett A, Armer-Cabral M, Marshall K, Kaur N, Bloom MS, Tabriziani H, Bhorade S, Cooper M; ProActive Investigators. Elevation of Donor-derived Cell-free DNA Before Biopsy-proven Rejection in Kidney Transplant. Transplantation. 2024 Sep 1;108(9):1994-2004. doi: 10.1097/TP.0000000000005007. Epub 2024 Aug 20. PMID 38595232